CLINICAL TRIAL: NCT00326898
Title: ASSURE: Adjuvant Sorafenib or Sunitinib for Unfavorable Renal Carcinoma
Brief Title: Sunitinib Malate or Sorafenib Tosylate in Treating Patients With Kidney Cancer That Was Removed By Surgery
Acronym: ASSURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Cancer and Leukemia Group B (Network); NCIC Clinical Trials Group (Network); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2009-00534; NCI-2009-00534 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CAN-NCIC-E2805; SWOG-E2805; ECOG-E2805; CDR0000478976; CALGB-E2805; E2805 (Other: ECOG-ACRIN Cancer Research Group); E2805 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2006-05-16; First posted 2006-05-17 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Clear Cell Renal Cell Carcinoma; Stage I Renal Cell Cancer AJCC v6 and v7; Stage II Renal Cell Cancer AJCC v7; Stage III Renal Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib; Sunitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (sunitinib malate, placebo) (Experimental): Beginning 4-12 weeks following radical or partial nephrectomy, patients receive sunitinib malate PO QD for 4 weeks and placebo sorafenib tosylate PO QD or BID for 6 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo; Other: Quality-of-Life Assessment; Drug: Sunitinib Malate
- Arm B (sorafenib tosylate, placebo) (Experimental): Beginning 4-12 weeks following radical or partial nephrectomy, patients receive sorafenib tosylate PO QD or BID for 6 weeks and placebo sunitinib malate PO QD for 4 weeks followed.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo; Other: Quality-of-Life Assessment; Drug: Sorafenib Tosylate
- Arm C (placebo) (Placebo Comparator): Beginning 4-12 weeks following radical or partial nephrectomy, patients receive placebo sorafenib tosylate as in Arm A and placebo sunitinib malate as in Arm B.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib
  Arms: Arm B (sorafenib tosylate, placebo)
Drug: Sunitinib Malate — Given PO
  Other Names: SU011248; SU11248; sunitinib; Sutent
  Arms: Arm A (sunitinib malate, placebo)

SUMMARY:
This randomized phase III trial studies sunitinib malate to see how well it works compared to sorafenib tosylate or placebo in treating patients with kidney cancer that has been removed by surgery. Sunitinib malate and sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving sunitinib malate or sorafenib tosylate after surgery may kill any tumor cells that remain after surgery. It is not yet known whether sunitinib malate is more effective than sorafenib tosylate or placebo in treating kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate an improvement in disease-free survival in locally advanced renal cell carcinoma patients randomly assigned to adjuvant sunitinib (sunitinib malate) (Arm A) or sorafenib (sorafenib tosylate) (Arm B) versus placebo (Arm C) after radical or partial nephrectomy.

SECONDARY OBJECTIVES:

I. To compare overall survival of patients randomized to each of the two regimens with placebo.

II. To further define the toxicity of prolonged administration of sunitinib or sorafenib in this patient population.

III. To prospectively collect tumor and biological specimens to assess their characteristics and associations: novel approaches to assess angiogenesis markers in tissue, blood and urine as predictors of disease-free survival and of therapeutic benefit.

IV. To prospectively collect tumor and biological specimens to assess their characteristics and associations: the frequency of oncogene and tumor suppressor gene mutations as predictors of disease-free survival and therapeutic benefit.

V. To prospectively collect tumor and biological specimens to assess their characteristics and associations: tumor and genetic polymorphisms as predictors of disease-free survival and therapeutic benefit.

VI. To prospectively collect tumor and biological specimens to assess their characteristics and associations: deoxyribonucleic acid (DNA) methylation profiles as predictors of outcome and of therapeutic benefit.

VII. To prospectively collect tumor and biological specimens to assess their characteristics and associations: The relationship of polymorphisms in drug metabolizing enzymes with steady state concentrations of sorafenib and sunitinib in selected patients.

VIII. To study the effect of vascular endothelial growth factor (VEGF) targeted therapy on circulating endothelial cells and circulating endothelial progenitors.

IX. To prospectively assess patient-reported fatigue in order to compare the magnitude and trajectory of fatigue among renal cell carcinoma (RCC) patients randomized to adjuvant sunitinib (Arm A) or sorafenib (Arm B) to placebo (Arm C). (Quality of life objectives) X. To evaluate the Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue-Short Form (SF)1, a newly developed state-of-the-science PROMIS measure for fatigue and to calibrate the PROMIS Fatigue-SF1 with the established, validated FACIT-Fatigue scale. (Quality of life objectives)

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM A: Beginning 4-12 weeks following radical or partial nephrectomy, patients receive sunitinib malate orally (PO) once daily (QD) for 4 weeks and placebo sorafenib tosylate PO QD or twice daily (BID) for 6 weeks.

ARM B: Beginning 4-12 weeks following radical or partial nephrectomy, patients receive sorafenib tosylate PO QD or BID for 6 weeks and placebo sunitinib malate PO QD for 4 weeks followed.

ARM C: Beginning 4-12 weeks following radical or partial nephrectomy, patients receive placebo sorafenib tosylate as in Arm A and placebo sunitinib malate as in Arm B.

In all arms, treatment repeats every 6 weeks for 9 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then every 12 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Pre-surgical criteria:

  * Patients must have primary-intact renal cell carcinoma, eligible for nephrectomy with curative intent
  * Tumors >= 4 cm AND/OR macroscopic fully resectable nodes AND/OR surgically resectable renal vein thrombus AND/OR surgically resectable inferior vena caval thrombus by radiologic criteria to be clinically >= pT1bNany (resectable) M0 disease
  * Multifocal ipsilateral renal cell carcinoma is allowed provided fully resectable and does not exceed inclusion criteria
* Patients must have no history of distant metastases
* No prior anti-cancer therapy for renal cell carcinoma is permitted in either the adjuvant or neoadjuvant setting; this includes metastectomy for renal cell carcinoma, or radiation therapy to the renal bed
* Patients must not have other current malignancies, other than basal cell skin cancer, squamous cell skin cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast; patients with other malignancies are eligible if they have been continuously disease-free for >= 5 years prior to the time of registration
* Patients must have no serious intercurrent illness including, but not limited to, the following: clinically significant cardiovascular disease (e.g. uncontrolled hypertension, myocardial infarction, unstable angina); New York Heart Association grade II or greater congestive heart failure; serious cardiac arrhythmia requiring medication; grade II or greater peripheral vascular disease; or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not have any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism
* Patient must not have ongoing ventricular cardiac dysrhythmias of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 grade >= 2; patients with a history of serious ventricular arrhythmia (ventricular tachycardia [VT] or ventricular fibrillation [VF] >= 3 beats in a row) are also excluded; additionally, patients with ongoing atrial fibrillation are not eligible
* Patients must have corrected QT (QTc) interval < 500 msec on baseline electrocardiogram (EKG)
* Patient must not have hypertension that cannot be controlled by medications (>= diastolic blood pressure 100 mm Hg despite optimal medical therapy)
* Patient must not have pre-existing thyroid abnormality with thyroid stimulating hormone that cannot be maintained in the normal range with medication
* If female, patient must not be pregnant or breastfeeding; all females of childbearing potential must have a blood test or urine study within 2 weeks prior to pre-registration to rule out pregnancy; if pre-registration occurs prior to surgery, the blood or urine study must be repeated within 2 weeks prior to randomization to rule out pregnancy; (note: should a woman become pregnant while participating in this study, she should inform her treating physician immediately)
* Women of child-bearing potential and men must agree to use an accepted and effective method of contraception prior to study entry and for the duration of study participation; should a woman become pregnant while participating in this study, she should inform her treating physician immediately; if a man impregnates a woman while participating in this study, he should inform his treating physician immediately as well
* Patients with known human immunodeficiency virus (HIV) are excluded
* ELIGIBILITY CRITERIA FOLLOWING RADICAL OR PARTIAL NEPHRECTOMY
* The date of randomization must be less than 12 weeks after the date of surgery; patients must have recovered from any surgical related complications
* Within 4 weeks prior to randomization, patients must meet preoperative eligibility requirements
* Patients must have histologically or cytologically confirmed renal cell carcinoma. Using 2002 (American Joint Committee on Cancer [AJCC] 6th edition) TNM Staging, patients must be one of the following:

  * pT1b G3-4 N0 (or pNX where clinically N0) M0
  * pT2 G (any) N0 (or pNX where clinically N0) M0
  * pT3 G (any) N0 (or pNX where clinically N0) M0
  * pT4 G (any) N0 (or pNX where clinically N0) M0 or
  * T (any) G (any) N+ (fully resected) M0

    * Patients with microvascular invasion of the renal vein of any grade or stage (as long as M0) are also eligible
    * Patients must have undergone a full surgical resection (radical nephrectomy or partial nephrectomy) by either open or laparoscopic technique; clinical evidence of lymph node positivity requires removal of all clinically positive nodes; surgeons should designate extent of node dissection; all surgical specimens must have negative margins; patients with positive renal vein margins are eligible unless there is invasion of the renal vein wall at the margin (provided no other margins are positive)
* Patients must not have collecting duct carcinomas or medullary carcinomas
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patients must have an absolute baseline left ventricular ejection fraction (LVEF) of >= 50% by multigated acquisition (MUGA) scan within 4 weeks prior to randomization
* Patients must have paraffin-embedded tumor specimen available for central core review of tumor histology and other correlative studies; tumor samples will be shipped as specified
* Patients must have no evidence of residual or metastatic renal cell cancer as documented on computed tomography (CT) scans of the chest, abdomen, and pelvis, all with oral and intravenous (IV) contrast (magnetic resonance imaging [MRI] scans of the abdomen and pelvis with gadolinium and a non-contrast CT of the chest may be substituted if patient is not able to have CT scans with intravenous contrast); patients unable to tolerate either gadolinium or IV contrast should not participate in this study (limitations to a patient's renal function should be taken into consideration when screening for this study)
* Scans must be obtained within 4 weeks of randomization; changes on these scans that are felt to be post surgical must be documented
* Patients without reported lymph nodes in the resected surgical specimen and a reported pathologic stage (post-nephrectomy) of pNX MUST undergo a post-operative contrast-enhanced CT scan (or MRI with gadolinium) within 4 weeks of randomization to document that there is no evidence of residual disease
* Patients must not be taking cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine or phenobarbital), St John's Wort, ketoconazole, dexamethasone, the dysrhythmic drugs (terfenadine, quinidine, procainamide, sotalol, probucol, bepridil, indapamide or flecainide), haloperidol, risperidone, rifampin, grapefruit, or grapefruit juice within two weeks of randomization and during the course of therapy; (medications are not prohibited unless listed above); topical and inhaled steroids are permitted
* Patients must not receive any other investigational anti-cancer agents during the period on study
* Patients must not have a serious intercurrent illness, including ongoing or active infection requiring parental antibiotics
* Absolute granulocyte count (AGC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Serum creatinine =< 2.0 x upper limit of normal (ULN) or calculated creatinine clearance (CrCl) >= 30 mL/min (neither drug is cleared by the kidney)
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) =< 2.5 x ULN
* Patients must be able to swallow pills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1943 (Actual)
Dates: Start 2006-04-24 (Actual); Primary Completion 2015-08-27 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi S Balzer-Haas, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (987):
- United States (966):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Providence Hospital, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Banner Thunderbird Medical Center, Glendale, Arizona
  - Banner-University Medical Center Phoenix, Phoenix, Arizona
  - Western Regional CCOP, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group-Rogers, Rogers, Arkansas
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Washington Hospital, Fremont, California
  - Saint Jude Medical Center, Fullerton, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - Saint Rose Hospital, Hayward, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Loma Linda Healthcare System, Loma Linda, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Community Hospital of Monterey Peninsula, Monterey, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Northridge Hospital Medical Center, Northridge, California
  - Sutter Cancer Research Consortium, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Shasta Regional Medical Center, Redding, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - University of California San Diego, San Diego, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Veterans Administration-San Diego Medical Center, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Northbay Cancer Center, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - University of Colorado, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Montrose Memorial Hospital, Montrose, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Danbury Hospital, Danbury, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Yale University, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Southwest Florida Regional Medical Center, Fort Myers, Florida
  - Florida Cancer Specialists-Gainesville Cancer Center, Gainesville, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - Cancer Centers of Central Florida PA, Leesburg, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - 21st Century Oncology-Orange Park, Orange Park, Florida
  - AdventHealth Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Portneuf Medical Center, Pocatello, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - AMITA Health Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Cottage, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - LaGrange Oncology Associates, Geneva, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Vigliotti, Antonio, P.G. M.D. (UIA Investigator), Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - DuPage Medical Group-Ogden, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Franciscan St. James Health-Olympia Fields Campus, Olympia Fields, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Edward H Kaplan MD and Associates, Skokie, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Richard L. Roudebush Veterans Affairs Medical Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Horizon Oncology Research LLC, Lafayette, Indiana
  - Premier Oncology Hematology Associates, Merrillville, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Cancer Care Institute, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, Waterloo, Iowa
  - MercyOne Waterloo Medical Center, Waterloo, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Hays Medical Center, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Shawnee Mission Medical Center-KCCC, Shawnee Mission, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Doctors Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - University Health-Conway, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Mercy Hospital, Portland, Maine
  - Maine Center for Cancer Medicine-Scarborough, Scarborough, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Maine General Medical Center-Thayer, Waterville, Maine
  - York Hospital, York Village, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Memorial Hospital at Easton - Shore Regional Cancer Center, Easton, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Steward Saint Elizabeth's Medical Center, Brighton, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Holy Family Hospital, Methuen, Massachusetts
  - Milford Regional Medical Center, Milford, Massachusetts
  - Berkshire Medical Center - Cancer Center, Pittsfield, Massachusetts
  - Commonwealth Hematology Oncology PC-Worcester, Worcester, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Beaumont Hospital ? Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Harris, John Gilbert MD (UIA Investigator), Alexandria, Minnesota
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Brainerd Medical Center Inc, Brainerd, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Etzell, Paul S MD (UIA Investigator), Fergus Falls, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Swenson, Wade II, MD (UIA Investigator), Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Adult and Pediatric Urology PLLP, Sartell, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Missouri Cancer Associates, Columbia, Missouri
  - Veterans Administration, Columbia, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Freeman Health System, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Deaconess Medical Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson-Tahoe Specialty Medical Center, Carson City, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Frisbie Hospital, Rochester, New Hampshire
  - Ocean Medical Center, Brick, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Mountainside Hospital, Montclair, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Christus Saint Vincent Regional Medical Center, Santa Fe, New Mexico
  - New York Oncology Hematology PC - Albany, Albany, New York
  - New York Oncology Hematology PC -Albany Medical Center, Albany, New York
  - New York Oncology Hematology PC - Amsterdam, Amsterdam, New York
  - Kings County Hospital, Brooklyn, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Veteran Affairs New York Harbor Healthcare System-Brooklyn Campus, Brooklyn, New York
  - Veterans Affairs Western New York Health Care System-Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Oncology Hematology PC - Clifton Park, Clifton Park, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Adirondack Cancer Center, Glens Falls, New York
  - Glens Falls Hospital, Glens Falls, New York
  - New York Oncology Hematology PC-Hudson, Hudson, New York
  - Northwell Health NCORP, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Orange Regional Medical Center, Middletown, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Union Square, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Nyack Hospital, Nyack, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - New York Oncology Hematology PC - Rexford, Rexford, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Oncology Hematology PC - Troy, Troy, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Mission Hospital Inc-Memorial Campus, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Mid-Columbia Medical Center/Celilo Cancer Center, The Dalles, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, DuBois, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Armstrong Center for Medicine and Health, Kittanning, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Central PA Hematology-Medical Oncology Associates PC, Lemoyne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Aria Health-Torresdale Campus, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Associates In Hematology Oncology PC-Upland, Upland, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Hematology and Oncology Associates of Rhode Island Inc, Cranston, Rhode Island
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Kent Hospital, Warwick, Rhode Island
  - AnMed Health Hospital, Anderson, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Jones Clinic, Germantown, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - East Tennessee Baptist Hospital-Mercy Health Partners, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Nashville Oncology Associates PC, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Texas Oncology-Austin North, Austin, Texas
  - Texas Oncology Seton Northwest, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Texas Health Presbyterian Hospital Dallas, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Dallas Oncology Consultants PA, Duncanville, Texas
  - The Center for Integrative Cancer Medicine, El Paso, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Baylor Saint Luke's Medical Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - The Methodist Hospital System, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - Texas Oncology-Seton Williamson, Round Rock, Texas
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Oncology- San Marcos, San Marcos, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Peninsula Cancer Institute-Gloucester, Gloucester, Virginia
  - Centra Lynchburg Hematology-Oncology Clinic Inc, Lynchburg, Virginia
  - Peninsula Cancer Institute-Newport News, Newport News, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Peninsula Cancer Institute-Williamsburg, Williamsburg, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Providence Holy Family Hospital, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Cancer Institutes of Washington PLLC, Yakima, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Fox Valley Hematology and Oncology SC-Appleton, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Cancer Care-Franklin, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Glendale, Glendale, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - UW Health Oncology-One South Park, Madison, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (20):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Clinical Research Unit at Vancouver Coastal Health Authority, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Grand River Regional Cancer Centre at Grand River Hospital, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Algoma District Cancer Program Sault Area Hospital, Sault Ste. Marie, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - PEI Cancer Treatment Centre-Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Bottinor WJ, Flamand Y, Haas NB, ONeill AM, DiPaola RS, Subramanian P, Cella D, Hundley WG, Wagner LI, Salsman JM, Ky B. Cardiovascular Implications of Vascular Endothelial Growth Factor Inhibition Among Adolescents/Young Adults in ECOG-ACRIN E2805. J Natl Compr Canc Netw. 2023 Jul;21(7):725-731.e1. doi: 10.6004/jnccn.2023.7018. PMID 37433436
- [Derived] Karam JA, Puligandla M, Flaherty KT, Uzzo RG, Matin SF, Pins MR, Wood CG, Kane C, Jewett MAS, Kim SE, Dutcher JP, DiPaola RS, Haas NB. Adjuvant therapy in patients with sarcomatoid renal cell carcinoma: post hoc analysis from Eastern Cooperative Oncology Group-American College of Radiology Imaging Network (ECOG-ACRIN) E2805. BJU Int. 2022 Jun;129(6):718-722. doi: 10.1111/bju.15587. Epub 2021 Sep 23. PMID 34480522
- [Derived] Murphy CC, Fullington HM, Gerber DE, Bowman IA, Puligandla M, Dutcher JP, DiPaola RS, Haas NB. Adherence to oral therapies among patients with renal cell carcinoma: Post hoc analysis of the ECOG-ACRIN E2805 trial. Cancer Med. 2021 Sep;10(17):5917-5924. doi: 10.1002/cam4.4140. Epub 2021 Aug 18. PMID 34405965
- [Derived] Jamil ML, Keeley J, Sood A, Dalela D, Arora S, Peabody JO, Trinh QD, Menon M, Rogers CG, Abdollah F. Long-term Risk of Recurrence in Surgically Treated Renal Cell Carcinoma: A Post Hoc Analysis of the Eastern Cooperative Oncology Group-American College of Radiology Imaging Network E2805 Trial Cohort. Eur Urol. 2020 Feb;77(2):277-281. doi: 10.1016/j.eururo.2019.10.028. Epub 2019 Nov 6. PMID 31703971
- [Derived] Buti S, Puligandla M, Bersanelli M, DiPaola RS, Manola J, Taguchi S, Haas NB. Validation of a new prognostic model to easily predict outcome in renal cell carcinoma: the GRANT score applied to the ASSURE trial population. Ann Oncol. 2017 Nov 1;28(11):2747-2753. doi: 10.1093/annonc/mdx492. PMID 28945839
- [Derived] Haas NB, Manola J, Dutcher JP, Flaherty KT, Uzzo RG, Atkins MB, DiPaola RS, Choueiri TK. Adjuvant Treatment for High-Risk Clear Cell Renal Cancer: Updated Results of a High-Risk Subset of the ASSURE Randomized Trial. JAMA Oncol. 2017 Sep 1;3(9):1249-1252. doi: 10.1001/jamaoncol.2017.0076. PMID 28278333
- [Derived] Haas NB, Manola J, Uzzo RG, Flaherty KT, Wood CG, Kane C, Jewett M, Dutcher JP, Atkins MB, Pins M, Wilding G, Cella D, Wagner L, Matin S, Kuzel TM, Sexton WJ, Wong YN, Choueiri TK, Pili R, Puzanov I, Kohli M, Stadler W, Carducci M, Coomes R, DiPaola RS. Adjuvant sunitinib or sorafenib for high-risk, non-metastatic renal-cell carcinoma (ECOG-ACRIN E2805): a double-blind, placebo-controlled, randomised, phase 3 trial. Lancet. 2016 May 14;387(10032):2008-16. doi: 10.1016/S0140-6736(16)00559-6. Epub 2016 Mar 9. PMID 26969090
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on April 24, 2006 and closed to accrual on September 1, 2010, after accrual of 1943 patients.
Groups:
- Arm A (Sunitinib + Sorafenib Placebo): Beginning 4-12 weeks following radical or partial nephrectomy, patients receive sunitinib malate 37.5mg PO QD for 4 weeks and placebo sorafenib tosylate 400mg PO QD or BID for 6 weeks.
- Arm B (Sorafenib + Sunitinib Placebo): Beginning 4-12 weeks following radical or partial nephrectomy, patients receive sorafenib tosylate 400mg PO QD or BID for 6 weeks and placebo sunitinib malate 37.5mg PO QD for 4 weeks followed.
- Arm C (Sunitinib Placebo + Sorafenib Placebo): Beginning 4-12 weeks following radical or partial nephrectomy, patients receive placebo sorafenib tosylate 400mg as in Arm A and placebo sunitinib malate 37.5mg as in Arm B.
Period: Overall Study
Arm/Group | Arm A (Sunitinib + Sorafenib Placebo) | Arm B (Sorafenib + Sunitinib Placebo) | Arm C (Sunitinib Placebo + Sorafenib Placebo)
Started | 647 | 649 | 647
Patients With Toxicity Data | 625 | 628 | 626
Patients With Clear Cell Histology | 542 | 540 | 540
Patients With >=1 Follow-up MUGA Scan | 513 | 510 | 580
Completed | 296 | 306 | 444
Not Completed | 351 | 343 | 203
Not completed — Disease progression | 52 | 54 | 102
Not completed — Adverse Event | 124 | 128 | 33
Not completed — Death | 2 | 0 | 0
Not completed — Withdrawal by Subject | 134 | 128 | 32
Not completed — Alternative therapy | 1 | 0 | 0
Not completed — Other complicating disease | 5 | 5 | 4
Not completed — Other/Missing/Unknown | 33 | 28 | 32

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Sunitinib + Sorafenib Placebo) | Arm B (Sorafenib + Sunitinib Placebo) | Arm C (Sunitinib Placebo + Sorafenib Placebo) | Total
Number analyzed (Participants) | 647 | 649 | 647 | 1943
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 489 | 507 | 500 | 1496
  >=65 years | 158 | 142 | 147 | 447
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218 | 212 | 204 | 634
  Male | 429 | 437 | 443 | 1309

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: Disease-free survival (DFS) is defined as time from randomization to recurrence, development of second primary cancer (except localized breast or prostate cancer or nonmelanoma skin cancer), or death from any cause. Patients who were alive without recurrence or qualifying second primary cancer were censored at the date of last disease evaluation.
Time Frame: Assessed every 3 months if patient is < 2 years from study entry; every 6 months if patient is 2 - 5 years from study entry; then annually if patient is 5 - 10 years from study entry
Population: All randomized patients
Measure: Median (97.5% Confidence Interval); unit: years
Arm/Group | Arm A (Sunitinib + Sorafenib Placebo) | Arm B (Sorafenib + Sunitinib Placebo) | Arm C (Sunitinib Placebo + Sorafenib Placebo)
Number analyzed (Participants) | 647 | 649 | 647
years | 5.8 [5.0 to NA] — The upper limit of the 97.5% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 6.1 [4.8 to NA] — The upper limit of the 97.5% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 6.6 [5.3 to 7.8]
Statistical Analysis 1: Comparison: Arm A (Sunitinib + Sorafenib Placebo) vs Arm C (Sunitinib Placebo + Sorafenib Placebo); Test type: Superiority or Other; p = 0.80, Stratified logrank test; Stratified logrank test was performed. Stratification factors include basis of risk group, histologic subtype, performance status and type of surgery; Hazard Ratio (HR) = 1.02, 97.5% CI 2-sided [0.85 to 1.23]
Statistical Analysis 2: Comparison: Arm B (Sorafenib + Sunitinib Placebo) vs Arm C (Sunitinib Placebo + Sorafenib Placebo); Test type: Superiority or Other; p = 0.72, Stratified logrank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.97, 97.5% CI 2-sided [0.80 to 1.17]

2. Secondary Outcome: 5-year Overall Survival Rate
Description: Overall survival is defined as the time from randomization to death from any cause. Patients without a date of death were censored at the date of last contact. Kaplan-Meier method was used to estimate 5-year survival rate.
Time Frame: Assessed every 3 months if patient is < 2 years from study entry; every 6 months if patient is 2 - 5 years from study entry
Population: All randomized patients
Measure: Number (97.5% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Sunitinib + Sorafenib Placebo) | Arm B (Sorafenib + Sunitinib Placebo) | Arm C (Sunitinib Placebo + Sorafenib Placebo)
Number analyzed (Participants) | 647 | 649 | 647
proportion of participants | 0.779 [0.741 to 0.819] | 0.805 [0.768 to 0.842] | 0.803 [0.767 to 0.840]
Statistical Analysis 1: Comparison: Arm A (Sunitinib + Sorafenib Placebo) vs Arm C (Sunitinib Placebo + Sorafenib Placebo); Test type: Superiority or Other; Hazard Ratio (HR) = 1.17, 97.5% CI 2-sided [0.90 to 1.52] — Hazard ratio was estimated using stratified proportional hazards model with Arm C (placebo arm) as the reference group
Statistical Analysis 2: Comparison: Arm B (Sorafenib + Sunitinib Placebo) vs Arm C (Sunitinib Placebo + Sorafenib Placebo); Test type: Superiority or Other; Hazard Ratio (HR) = 0.98, 97.5% CI 2-sided [0.75 to 1.28] — Hazard ratio was estimated using stratified proportional hazards model with Arm C (placebo arm) as the reference group

3. Secondary Outcome: Proportion of Patients With Cardiac Events
Description: Cardiac event is defined as left ventricular ejection fraction (LVEF) below the institutional lower limit of normal, where the decrease was >15% absolute percentage points from baseline within 6 months.
Time Frame: as for outcome 2
Population: Patients with at least 1 follow-up MUGA scan were included in this analysis.
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A (Sunitinib + Sorafenib Placebo) | Arm B (Sorafenib + Sunitinib Placebo) | Arm C (Sunitinib Placebo + Sorafenib Placebo)
Number analyzed (Participants) | 513 | 510 | 580
Proportion of participants | 0.017 [0.009 to 0.030] | 0.013 [0.006 to 0.026] | 0.008 [0.003 to 0.018]

4. Secondary Outcome: 5-year Disease-free Survival (DFS) Rate Among Patients With Clear Cell Histology
Description: Disease-free survival (DFS) is defined as time from randomization to recurrence, development of second primary cancer (except localized breast or prostate cancer or nonmelanoma skin cancer), or death from any cause. Patients who were alive without recurrence or qualifying second primary cancer were censored at the date of last disease evaluation. 5-year DFS rate is the proportion of patients who are alive and disease-free at 5 years based on the Kaplan-Meier estimate.
Time Frame: as for outcome 1
Population: Patients with clear cell histology were included in this analysis.
Measure: Number (97.5% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Sunitinib + Sorafenib Placebo) | Arm B (Sorafenib + Sunitinib Placebo) | Arm C (Sunitinib Placebo + Sorafenib Placebo)
Number analyzed (Participants) | 542 | 540 | 540
proportion of participants | 0.534 [0.484 to 0.590] | 0.527 [0.478 to 0.582] | 0.560 [0.511 to 0.614]

5. Other Pre Specified Outcome: The Association Between Angiogenesis Markers and Disease-free Survival
Time Frame: as for outcome 1
Reporting Status: Not Posted

6. Other Pre Specified Outcome: The Association Between Disease-free Survival and the Frequency of Oncogene as Well as Tumor Suppressor Gene Mutations
Time Frame: as for outcome 1
Reporting Status: Not Posted

7. Other Pre Specified Outcome: The Association Between Tumor and Genetic Polymorphisms and Disease-free Survival
Time Frame: as for outcome 1
Reporting Status: Not Posted

8. Other Pre Specified Outcome: The Association Between Deoxyribonucleic Acid (DNA) Methylation Profiles and Disease-free Survival
Time Frame: as for outcome 1
Reporting Status: Not Posted

9. Other Pre Specified Outcome: The Relationship of Polymorphisms in Drug Metabolizing Enzymes With Steady State Concentrations of Sorafenib and Sunitinib in Selected Patients
Time Frame: as for outcome 1
Reporting Status: Not Posted

10. Other Pre Specified Outcome: The Effect of Vascular Endothelial Growth Factor (VEGF) Targeted Therapy on Circulating Endothelial Cells and Circulating Endothelial Progenitors
Time Frame: as for outcome 1
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Patient-reported Fatigue Using Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue Scale
Time Frame: Assessed at baseline, 10 weeks and 22 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Patient-reported Fatigue Using the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form
Description: PROMIS Fatigue short form is a newly developed state-of-the-science PROMIS measure for fatigue
Time Frame: Assessed at baseline, 10 weeks and 22 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: The Association Between Scan Frequency and Development of Congestive Heart Failure
Time Frame: Assessed at 3, 6 and 12 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Frequency of Clinically Significant Congestive Heart Failure (CHF) Grade 3 or Higher Using the Common Terminology Criteria for Adverse Events Version 4.0
Time Frame: Assessed every 6 weeks while on treatment and for 30 days after the end of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 6 weeks while on treatment and for 30 days after the end of treatment
Description: Only adverse events that are possibly, probably, or definitely related to protocol therapy are reported.
Arm/Group | Arm A (Sunitinib + Sorafenib Placebo) | Arm B (Sorafenib + Sunitinib Placebo) | Arm C (Sunitinib Placebo + Sorafenib Placebo)
Serious Adverse Events (participants affected / at risk) | 368/625 | 424/628 | 81/626
Other Adverse Events (participants affected / at risk) | 116/625 | 117/628 | 57/626
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Sunitinib + Sorafenib Placebo) (N=625) | Arm B (Sorafenib + Sunitinib Placebo) (N=628) | Arm C (Sunitinib Placebo + Sorafenib Placebo) (N=626)
Allergic reaction (Immune system disorders) | 1 | 0 | 0
Hearing w/o audiogr not in monitor prg (Ear and labyrinth disorders) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 1 | 0
Leukocytes decreased (Investigations) | 3 | 0 | 0
Neutrophils decreased (Investigations) | 7 | 2 | 0
Platelets decreased (Investigations) | 13 | 2 | 1
Heart block abnormality NOS (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 0 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Vasovagal episode (Nervous system disorders) | 1 | 0 | 0
Bigeminy (Cardiac disorders) | 1 | 0 | 0
Cardiac-ischemia (Cardiac disorders) | 1 | 3 | 4
Hypertension (Vascular disorders) | 104 | 96 | 15
Hypotension (Vascular disorders) | 1 | 0 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 4 | 4 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cor Pulmonale (Cardiac disorders) | 0 | 1 | 0
cardiac-other (Cardiac disorders) | 0 | 1 | 0
Fatigue (General disorders) | 108 | 41 | 15
Fever w/o neutropenia (General disorders) | 1 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 4 | 0
Weight gain (Investigations) | 0 | 0 | 2
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 | 11 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 15 | 93 | 3
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 94 | 208 | 7
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Wound - non-infectious (Injury, poisoning and procedural complications) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Hyopthyroidism (Endocrine disorders) | 2 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 11 | 5 | 0
Colitis (Gastrointestinal disorders) | 0 | 3 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 10 | 3 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 57 | 55 | 2
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 14 | 4 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 2 | 0 | 0
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 3 | 1 | 0
Muco/stomatitis (symptom) pharynx (Respiratory, thoracic and mediastinal disorders) | 24 | 14 | 0
Nausea (Gastrointestinal disorders) | 22 | 5 | 0
Perforation, colon (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 11 | 3 | 1
Colon, hemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Lower GI, hemorrhage NOS (Gastrointestinal disorders) | 0 | 1 | 0
Stomach, hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Kidney, hemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Liver dysfunction/failure (Hepatobiliary disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 1 | 0
Hepatic-other (Hepatobiliary disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Infection w/ gr3-4 neut, ileum (Infections and infestations) | 1 | 0 | 0
Infection Gr0-2 neut, appendix (Infections and infestations) | 0 | 0 | 1
Infection Gr0-2 neut, colon (Infections and infestations) | 0 | 2 | 0
Infection Gr0-2 neut, kidney (Infections and infestations) | 1 | 1 | 0
Infection Gr0-2 neut, lung (Infections and infestations) | 2 | 3 | 2
Infection Gr0-2 neut, mediastinm (Infections and infestations) | 0 | 0 | 1
Infection Gr0-2 neut, mucosa (Infections and infestations) | 0 | 1 | 0
Infection Gr0-2 neut, muscle (Infections and infestations) | 0 | 1 | 0
Infection Gr0-2 neut, nerve-cranial (Infections and infestations) | 1 | 0 | 0
Infection Gr0-2 neut, skin (Infections and infestations) | 0 | 1 | 0
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 1 | 0 | 1
Infection Gr0-2 neut, vagina (Infections and infestations) | 1 | 0 | 0
Infection Gr0-2 neut, wound (Infections and infestations) | 0 | 1 | 0
Infection w/ unk ANC skin (cellulitis) (Infections and infestations) | 0 | 2 | 0
Infection w/ unk ANC urinary tract NOS (Infections and infestations) | 0 | 1 | 0
Infection Gr0-2 neut, blood (Infections and infestations) | 1 | 0 | 0
Infection-other (Infections and infestations) | 1 | 1 | 0
Edema head and neck (General disorders) | 3 | 1 | 0
Edema limb (General disorders) | 2 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 4 | 0
Serum amylase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 6 | 4 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypercholesterolemia (Investigations) | 1 | 0 | 0
CPK increased (Investigations) | 1 | 1 | 0
Creatinine increased (Investigations) | 1 | 3 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Lipase increased (Investigations) | 4 | 3 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 2 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 5 | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 3
Nonneuropathic upper extr muscle weak (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Nonneuropathic left-side muscle weak (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nonneuropathic right-side muscle weak (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 4 | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 0
Confusion (Psychiatric disorders) | 2 | 0 | 1
Dizziness (Nervous system disorders) | 4 | 2 | 2
Memory impairment (Nervous system disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 2 | 2
Neuropathy-motor (Nervous system disorders) | 3 | 1 | 0
Neuropathy-sensory (Nervous system disorders) | 3 | 12 | 3
Syncope (Nervous system disorders) | 4 | 2 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Double vision (Eye disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 0
Ocular-other (Eye disorders) | 0 | 1 | 0
Abdomen, pain (Gastrointestinal disorders) | 4 | 8 | 2
Back, pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Bone, pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Cardiac/heart, pain (Cardiac disorders) | 2 | 3 | 0
Chest/thoracic pain NOS (General disorders) | 4 | 4 | 0
Esophagus, pain (Gastrointestinal disorders) | 1 | 0 | 0
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0
Head/headache (Nervous system disorders) | 6 | 4 | 0
Joint, pain (Musculoskeletal and connective tissue disorders) | 8 | 8 | 3
Muscle, pain (Musculoskeletal and connective tissue disorders) | 2 | 8 | 1
Oral cavity, pain (Gastrointestinal disorders) | 1 | 1 | 0
Scalp, pain (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Skin, pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Stomach, pain (Gastrointestinal disorders) | 0 | 1 | 0
Pain-other (General disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 2
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 6 | 4 | 0
Renal/GU-other (Renal and urinary disorders) | 0 | 1 | 0
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Sexual/Reproductive function-Other (Reproductive system and breast disorders) | 0 | 1 | 0
Flu-like syndrome (General disorders) | 3 | 0 | 0
Vascular access,Thrombosis/embolism (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 3 | 5 | 1
Vascular-Other (Specify) (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Sunitinib + Sorafenib Placebo) (N=625) | Arm B (Sorafenib + Sunitinib Placebo) (N=628) | Arm C (Sunitinib Placebo + Sorafenib Placebo) (N=626)
Hypertension (Vascular disorders) | 38 | 38 | 10
Fatigue (General disorders) | 62 | 58 | 31
Rash/desquamation (Skin and subcutaneous tissue disorders) | 17 | 43 | 15
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 36 | 52 | 7
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 41 | 40 | 13
Nausea (Gastrointestinal disorders) | 33 | 21 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less